CLINICAL TRIAL: NCT06392828
Title: EndoNAFLD: Evaluation of the Relationship Between Fatty Liver Disease and Endothelial Damage in Patients at High Risk of Cardiovascular Disease
Brief Title: EndoNAFLD: Relationship Between Fatty Liver Disease and Cardiovascular Diseases
Acronym: Endo-NAFLD
Status: Recruiting | Type: Observational
Sponsor: IMDEA Food (Other)
Collaborators: Sociedad Española de Arteriosclerosis (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital HM Montepríncipe (Unknown); Hospital Central de la Defensa Gómez Ulla (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Lidia Daimiel Ruiz, Principal Investigator, IMDEA Food
Other Study IDs: PI-058
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Cardiovascular Diseases
Keywords: endothelial damage; microbiota; liver disease; fatty liver disease; NAFLD; MAFLD; cardiovascular disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, PBMCs, urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: no NAFLD, no prevalent CVD.: The aim of this group is to serve as control group. FLI <30 or hepatic echography negative for liver steatosis if FLI >30; FLI < 60, con SCORE2 < 5 % and no prevalent CVD according to ESC 202122.
- Group 2: NAFLD, no prevalent CVD: FLI >60 or hepatic echography positive for liver steatosis if FLI >30; FLI < 60, con SCORE2 > 5 % and no prevalent CVD according to ESC 202122.
- Group 3: no NAFLD, prevalent CVD: FLI <30 or hepatic echography negative for liver steatosis if FLI >30; FLI < 60, con SCORE2 < 5 % and prevalent CVD (chest angina, stroke, acute coronary syndrome, accute myocardial infarction).
- Group 4: NAFLD, prevalent CVD: FLI >60 or hepatic echography positive for liver steatosis if FLI >30; FLI < 60, con SCORE2 > 5 % and prevalent CVD (chest angina, stroke, acute coronary syndrome, accute myocardial infarction).

SUMMARY:
Management of risk factors is the primary approach to prevent cardiovascular disease (CVD). In this regard the accurate scoring of disease risk is fundamental. Non-alcoholic fatty liver disease (NAFLD) has emerged recently as a potential mediator of CVD onset and progression. The hypothesis is that NAFLD can be a predictive CVD risk factor, independent of other classical and well-known risk factors.

Preliminary epidemiological studies suggested that the fat infiltration in the liver mirrored the cardiometabolic status of the patient. But recent studies postulate that NAFLD could be a potential independent predictor of vascular injury.

The mechanisms that link liver function and endothelial damage include modulation of adipose tissue function, lipid metabolism regulation or glycemic homeostasis, among others. But new mechanisms that could link NAFLD and ECV are emerging. The synthesis of ketone bodies in the liver is closely related to the cardiovascular system function. Ketone bodies can provide up to 50% of energy required by specific tissues. Plasma concentration of β-hydroxybutyrate is a biomarker of NAFLD. Plasma β-hydroxybutyrate and acetoacetate levels are also inversely associated with endothelial injury.

Other biomarkers on endothelial damage like von Willebrand factor, ICAM, VCAM or coagulation factors (Factor VIII) can be used to stratify patients according to the risk of CVD. The improvement in the sensitivity, specificity and accuracy of scores such as FLI, HIS and FIB-4 and non-invasive techniques such as elastography allow the study of the relationship between liver disease and other comorbidities.

The aim is to evaluate the potential of NAFLD to stratify patients according to the risk of CVD and to investigate the molecular mechanisms linking NAFLD and CVD.

DETAILED DESCRIPTION:
The hypothesis is that the prevalence of NAFLD and its degree, evaluated with non-invasive techniques and biomarkers is an independent risk factor of cardiovascular disease and can be used in scoring systems to stratify patients according to CVD risk.

The specific objectives are:

O1) To define the association between NAFLD prevalence and degree and endothelial damage.

The investigators will use non-invasive methods to determine the presence and degree of NAFLD (FLI, echography, elastography, FIB-4, NAFLD score and Hepamet) and the investigators will compare plasma concentrations of endothelial damage biomarkers (Von Willebrand Factor, Factor VIII and Tissue Factor) among NAFLD degrees.

O2) To describe the role of hepatic ketogenic metabolism as mediator of endothelial damage.

The investigators will correlate plasma concentrations of β-hydroxybutyrate and keto acetone with plasma concentrations of biomarkers of endothelial damage.

O3) To compare the expression of genes and microRNAs involved in endothelial function and liver metabolism and inflammation biomarkers among groups.

Liver metabolism is strictly regulated through the regulation of the expression of genes encoding metabolic enzymes responsible for the metabolic reactions and transporters of intermediate metabolites. The expression of such genes also depends on epigenetic mechanisms like microRNAs. Thus, the investigators will compare the expression of a selected panel of genes and microRNAs in blood samples of participants according to the clinicopathological group. The investigators will measure circulating microRNAs in plasma and cellular genes and microRNAs in the cellular fraction of the blood samples.

O4) To determine the role of the microbiome as mediator of the link between NAFLD and CVD.

The investigators will collect fecal samples from participants, and the investigators will compare alpha diversity and composition of the gut microbiota of the volunteers of the different clinicopathological groups. The investigators will also carry out comparative metagenomic studies.

Objectives 1 to 4 will be developed through a cross-sectional study in the participants.

O5) To associate NAFLD with the incidence of CVD events or changes in endothelial damage biomarkers.

Recruited participants with or without prevalent CVD will be followed up for 5 years to evaluate if the prevalence of NAFLD is associated with the incidence of CVD major events (cardiovascular mortality, myocardial infarction, stroke or chest angina).

To develop this aim, the investigators will carry out a longitudinal cohort study for 5 years. Participants recruited in any of the 4 clinicopathological groups will be contacted annually for 5 years to collect clinical, lifestyle and anthropometrical data. They will be also submitted to usual care protocols for their pathologies. Clinical records will be checked to assess the incidence of CVD events.

The aim is to recruit 112 participants, men and women, 50-69 years old that will be segregated according to NAFLD and CVD status:

Group 1: no NAFLD, no prevalent CVD. Group 2: NAFLD, no prevalent CVD Group 3: no NAFLD, prevalent CVD Group 4: NAFLD, prevalent CVD No NAFLD is described as Fatty Liver Index (FLI) <30 or hepatic echography negative for liver steatosis if FLI >30 or FLI < 60, con SCORE2 < 5 %.

NAFLD is described as FLI > 60 or hepatic echography positive for liver steatosis if FLA>30 or FLI < 60, con SCORE2 > 5 %.

Prevalent CVD is defined according to ESC 2011 guidelines (chest angina, stroke, acute coronary syndrome or acute myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 50-69 years old
* With CVD stratification according to ESC 2011 guidelines.
* With data to calculate NAFLD scores.

Exclusion Criteria:

Exclusion Criteria:

* Type 1 or type 2 diabetes.
* Taking hypoglycemic drugs.
* Familiar hypercholesterolemia according to ESC criteria.
* Congenital defects on lipid metabolism.
* Taking hypolipidemic drugs targeting PCSK9.
* Participating on other clinical trials.
* Chronic renal disease with filtration rate < 30 ml/min (RCD degree 4 KDIGO).
* Active cancer
* Liver disease no NAFLD.
* Von Willebrand disease or any other genetic condition with an impact on the plasma concentration of this biomarker.
* Systemic autoimmune disease.
* Uncapable of giving informed consent.
* Any other physical or cognitive condition that could affect the participation in the study.

Ages: 50 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending internal medicine services from the collaborating hospitals will be invited to participate. Physicians responsible for their usual care will check inclusion/exclusion criteria before inviting them to participate.
  All participants are community-dwelling adults from Community of Madrid, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endothelial damage | 5 years
  Measure of plasma concentration of Von Willebrand Factor in UI/dL
Endothelial damage | 5 years
  Measure of plasma concentration of Factor VIII in UI/mL
Endothelial damage | 5 years
  Measure of plasma concentration of Tissue Factor in ng/mL

SECONDARY OUTCOMES:
Endothelial dysfunction | 5 years
  Measure of plasma concentration of ICAM and VCAM measured, both, in ng/mL
Inflammatory status | 5 years
  Measure of plasma concentration of TNF-alpha, IL-1B and IL-6, measured in ng/mL
Ketogenic metabolism | 5 years
  Measure of blood levels of beta-hydroxybutyrate
Genomic profile | 5 years
  Measure of the relative expression, through Real-Time qPCR, of a panel of selected genes.
MicroRNA profile | 5 years
  Measure of the relative expression, through Real-Time qPCR, of a panel of selected microRNAs.
Microbiota diversity | 5 years
  Measure of alpha diversity and gut microbial composition through 16S sequencing of fecal samples.
Microbiota functionality | 5 years
  Metagenomic analysis of microbiota genes by sequencing
Cardiovascular disease incidence | 5 years
  Registration of major cardiovascular events (cardiovascular mortality, chest angina, accute myocardial infarction and stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Daimiel Ruiz, PhD, Principal Investigator — Fundación IMDEA Alimentación; Diego Martínez Urbistondo, PhD, Study Chair — Clínica Universidad de Navarra
Locations (4):
- Spain (4):
  - Clínica Universidad de Navarra, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Central de la Defensa Gomez Ulla, Madrid
  - Hospital HM Montepríncipe, Madrid

IPD SHARING:
Plan to Share IPD: No
IPD will no be available for other researchers. Study database can be accessible totally or partially upon request to study coordinator.